CLINICAL TRIAL: NCT03892070
Title: Beta-Hydroxy-Beta-Methylbutyrate Supplementation and Physical Activity in Liver Cirrhosis: a Controlled Trial
Acronym: HMB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Manuela Merli, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5038
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Sarcopenia; Cirrhosis, Liver
Keywords: HMB; Physical exercise
MeSH Terms: conditions — Sarcopenia; Liver Cirrhosis; Motor Activity | interventions — beta-hydroxyisovaleric acid; Mannitol

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: patients do not know if they are placebo or HMB group. Investigators who perform measurement and patients visit do not know the group of patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMB GROUP (Experimental): HMB Supplementation with 1.5 g of HMB taken twice daily. Supplementation will be provided for 12 weeks
  Interventions: Dietary Supplement: BETA-HYDROXY-BETA-METHYLBUTYRATE (HMB)
- PLACEBO GROUP (Placebo Comparator): Mannitol 1.5 g twice daily. Supplementation will be provided for 12 weeks
  Interventions: Dietary Supplement: Mannitol

INTERVENTIONS:
Dietary Supplement: BETA-HYDROXY-BETA-METHYLBUTYRATE (HMB) — 1.5 g of HMB will be provided for 12 weeks twice daily
  Arms: HMB GROUP
Dietary Supplement: Mannitol — 1.5 g twice daily for 12 weeks
  Arms: PLACEBO GROUP

SUMMARY:
Sarcopenia is an independent predictor of morbidity and mortality in the cirrhotic patient. Beta-hydroxy-beta-methyl butyrate (HMB) is a leucine metabolite with potential efficacy in increasing protein synthesis, muscle mass, and its functionality.

The aim of this randomized controlled study is to evaluate the effect of nutritional supplementation with HMB and physical activity both on muscle mass and on muscle function in cirrhotic patients.

DETAILED DESCRIPTION:
1. Introduction Changes in nutritional status are a frequent complication in cirrhotic patients. The prevalence of malnutrition is related to the severity of the disease and has been reported by 65-90% in advanced cirrhosis. The most significant component of malnutrition is a progressive and generalized loss of mass understood as sarcopenia.

   Several studies have reported that sarcopenia represents a negative prognostic factor for survival in patients with liver cirrhosis. Other studies have shown that sarcopenia is an independent predictor of complications of portal hypertension.

   For these reasons and being a modifiable condition, identifying and treating sarcopenia in patients is very important for their prognosis.

   Sarcopenia in liver cirrhosis occurs as a result of an increase in proteolysis or a reduction in protein synthesis, or a combination of the two mechanisms. The alterations in the molecular pathways that involve the regulation of these mechanisms are not entirely known. Recent research has led to the identification of increased expression of myostatin, member of the transforming growth factor ß superfamily, in skeletal muscle in animal models of hepatic injury and in the plasma of cirrhotic patients with consequent inhibition of protein synthesis. In addition, myostatin is able to examine the protein kinase 5' AMP-activated protein kinase (AMPK), an inhibitor of signaling of mammalian target of rapamycin (mTOR), a key regulator of protein synthesis.

   I populations of non-cirrhotic malnourished patients, the benefits of a therapy aimed at improving malnutrition are highlighted by reduced mortality, infections, systemic inflammatory responses and hospital stay. For cirrhotic patients, specific studies in this regard are limited by the size of the cohort and by the design of the study, and there are no effective therapies mainly due to the fact that the mechanisms of muscle loss in cirrhosis are not yet well understood. In addition, the end-points of these studies are heterogeneous (regain muscle strength, the disappearance of sarcopenia, mortality, complications of portal hypertension, etc.). In a study that used a nutritional enteral supplement, the authors observed a modest improvement in nutritional parameters but found no statistically significant differences in morbidity and mortality between the two patient groups. Better results have been reported in clinical trials that used nocturnal nutritional support, in most cases represented by branched-chain amino acids (BCAA) (leucine, isoleucine, and valine). This type of intervention has obtained an improvement in the use of energy substrates in the short term and an improvement of some nutritional parameters in the long term.

   Beta hydroxy-beta-methyl-butyrate (HMB) is a leucine metabolite with the potential to increase muscle performance and tropism. Studies conducted in experimental models of cachexia have reported increased phosphorylation and activation of mTOR secondary to the use of HMB. Experimental studies performed on cell cultures of myoblasts also showed an increased expression of insulin like growth factor-1 (IGF-1) secondary to treatment with HMB. These findings confirm the anabolic properties of HMB. A role of HMB on the suppression of proteolysis by inhibiting the ubiquitin-proteasome pathway in models of neoplastic cachexia and an effect on attenuating muscle atrophy secondary to steroid therapy has also been demonstrated. The association of anabolic properties targeting mTOR and anti-proteolytic make HMB a potential efficacy supplement for the treatment of sarcopenia in the cirrhotic patient. There are currently no data in the literature on the use of HMB in this category of patients.
2. Aim of the study

   Primary endpoints:

   • evaluate the effect at 3 months (T12) of HMB supplementation for 12 weeks in patients with liver cirrhosis on the mass and muscle performance compared to a group of patients

   The secondary objectives are:
   * assessment of the impact of supplementation with HMB on the development of complications (minimal and manifest hepatic encephalopathy, bacterial infections, ascites, GI bleeding) compared to the control group;
   * evaluation of the impact of sarcopenia on the number of admissions and the days of hospitalization for these complications compared to the control group;
   * identification of surrogate markers of sarcopenia through the preparation of a serum;

   This controlled trial is not sponsored by a drug company.
3. Patients Patients are enrolled in the study after been informed of the purpose and protocol of treatment and need to sign a written informed consent.
4. Statistical analysis, sample size, and randomization:

   For categorical variables, the Person-Chi-square test or the Fischer test will be used. For continuous variables, the Mann-Whitney Test will be used. The ANOVA variance analysis will be applied followed by the "t-test" when significant differences will be highlighted. Values of p <0.05 will be considered statistically significant.

   Block randomization, consisting of 4 individuals per block, was executed in a 1:1ratio using random numbers generated by an independent statistician (SPSS version 16.0). Knowledge of the randomization code was limited to the physician.

   While there is no evidence of HMB supplementation in cirrhotic patients, based on previously described variations in muscle mass in the elderly population, we aim to conduct a pilot study in which will be enrolled 20 patients per group.
5. Protocol of the study:

The registration will include the main clinical and biochemical data of patients.

Nutritional counseling will be provided to all patients to ensure similar caloric and daily protein intake in the two groups, according to the current guidelines (caloric intake of 20-25 kcal/kg/ die ± 10%, protein intake of 1.2 g /kg/day).

At the time of the enrollment and during the subsequent controls the following data will be recorded :

* calorie intake in the week preceding the visit by a three days non-consecutive food diary;
* height, weight, body mass index
* body composition by bioelectrical impedance analysis bioimmunoassay (BIA)
* muscular function evaluated by 6-minute walk test (6MWT), Timed Up and Go test-TUGT), e l'Hand grip Test (HG).
* biochemical and metabolic parameters
* pharmacological therapy During the study, clinical complications (hospital admissions, infectious events, the onset of comorbidity) will be recorded.

During the study, the tolerability of the supplement (analog-visual scale), adherence to absorption and any intolerance or secondary adverse effects will be detected.

Randomization: Patients are randomized to Group 1 - placebo (or control group) and Group 2 - supplementation (or treatment group)

The placebo will be 1gr mannitol twice daily. Supplementation will be HMB 1.5 g dissolved twice daily. Supplementation/placebo will be provided for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* all cirrhotics followed in outpatients' clinic 18-70 years

Exclusion Criteria:

* hepatocellular carcinoma or other neoplastic diseases;
* neuromuscular or skeletal diseases,
* chronic renal failure II-III degree;
* cardiac decompensation with New York Heart Association (NYHA) score ≥ III;
* severe pulmonary dysfunction;
* active alcohol intake in the last 6 months;
* ascites grade moderate-severe

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-10 (Estimated); Study Completion 2020-09-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Fat Free Mass Index after 12 weeks of supplementation | 12 weeks after the enrollment
  Increase of Fat Free Mass evaluated by BIA

SECONDARY OUTCOMES:
Changes in Fat Free Mass Index after 24 weeks of supplementation | 24 weeks after the enrollment
  Increase of Fat Free Mass evaluated by BIA
Changes in HG Test at 12 and 24 weeks after enrollment | 12 and 24 weeks after enrollment
  Recovery of muscle mass function evaluated by Recovery of muscle mass function evaluated by Hand grip Test (HG)
Changes in 6MWT Test at 12 and 24 weeks after enrollment | 12 and 24 weeks after enrollment
  Recovery of muscle mass function evaluated by 6 minute walk test-6MWT
Evaluation og Animal Naming and The Psychometric Hepatic Encephalopathy Score (PHES) | 12 and 24 weeks after enrollment
  evaluation of minimal hepatic encephalopathy
Evaluation of hospitalization and decompensation episodes | 12 and 24 weeks after enrollment
  episodes of decompensation during th study

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Department, Sapienza University of Rome, Rome, Italy

REFERENCES:
- [Background] Giusto M, Lattanzi B, Albanese C, Galtieri A, Farcomeni A, Giannelli V, Lucidi C, Di Martino M, Catalano C, Merli M. Sarcopenia in liver cirrhosis: the role of computed tomography scan for the assessment of muscle mass compared with dual-energy X-ray absorptiometry and anthropometry. Eur J Gastroenterol Hepatol. 2015 Mar;27(3):328-34. doi: 10.1097/MEG.0000000000000274. PMID 25569567
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Montano-Loza AJ, Meza-Junco J, Prado CM, Lieffers JR, Baracos VE, Bain VG, Sawyer MB. Muscle wasting is associated with mortality in patients with cirrhosis. Clin Gastroenterol Hepatol. 2012 Feb;10(2):166-73, 173.e1. doi: 10.1016/j.cgh.2011.08.028. Epub 2011 Sep 3. PMID 21893129
- [Background] Molfino A, Gioia G, Rossi Fanelli F, Muscaritoli M. Beta-hydroxy-beta-methylbutyrate supplementation in health and disease: a systematic review of randomized trials. Amino Acids. 2013 Dec;45(6):1273-92. doi: 10.1007/s00726-013-1592-z. Epub 2013 Sep 22. PMID 24057808
- [Background] Aversa Z, Alamdari N, Castillero E, Muscaritoli M, Rossi Fanelli F, Hasselgren PO. beta-Hydroxy-beta-methylbutyrate (HMB) prevents dexamethasone-induced myotube atrophy. Biochem Biophys Res Commun. 2012 Jul 13;423(4):739-43. doi: 10.1016/j.bbrc.2012.06.029. Epub 2012 Jun 13. PMID 22705301